CLINICAL TRIAL: NCT05505695
Title: The Effect of Schroth Exercises on Pulmonary Function in Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Halic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Schroth Exercises
Record Dates: First submitted 2022-07-30; First posted 2022-08-18 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-07

CONDITIONS: Adolescent Idiopathic Scoliosis; Pulmonary Function
MeSH Terms: interventions — Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Brace&Exercise Group" (Experimental): The patients who were the rigid brace and performed the SSE therapy in the specified constituted the Brace & Exercise. Experimental group patients wore full-time rigid brace and Schroth exercises for 60 minutes 5 days a week by the physician.
  Interventions: Other: Brace and Exercise Treatment
- "Brace Group" (Active Comparator): The patients who wore full-time rigid braces but did not perform exercise constituted the Brace group. Comparator group patients wore full-time brace only, did not perform Schroth exercises.
  Interventions: Other: Brace Treatment

INTERVENTIONS:
Other: Brace and Exercise Treatment — Schroth exercises, which are a specific exercise method for scoliosis, were given to the experimental group for 8 weeks, different from the control group.
  Arms: "Brace&Exercise Group"
Other: Brace Treatment — Among the patients included in the study, those who wore braces but did not agree to exercise constituted the ''Brace Group'' of the study.
  Arms: "Brace Group"

SUMMARY:
Background: In the present study, we aimed to evaluate the effect of regular Schroth exercises on pulmonary functions in adolescent idiopathic scoliosis (AIS) patients who use rigid braces and perform Schroth exercises regularly.

Objective: The main purpose of this study, is to investigate the effects of Schroth exercises on pulmonary functions in adolescents who use rigid braces and perform Schroth exercises regularly.

Methods: Twenty-four patients with AIS were included in the study. The patients who wore rigid braces and performed the SSE therapy constituted the "Brace&Exercise" (N=12), and the patients who wore full-time rigid braces but did not perform exercise constituted the "Brace Group" (N=12) of the study. The effects of Schroth exercises on pulmonary functions were measured at the beginning of treatment and the 8th week of the treatment.

Keywords: Adolescent, idiopathic scoliosis, conservative treatment, brace, respiratory function, Schroth exercises.

ELIGIBILITY:
Inclusion Criteria:

* 10-16 years,
* 25-45 Cobb degree,
* Brace and exercise treatment prescribed by the physician
* Participation in the study was approved by the family/caregiver

Exclusion Criteria:

* Chronic respiratory diseases,
* Professional athletes,
* Did not perform the exercises regularly
* Did not compliance the brace

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
FVC - Respiratory Functions | 8 Weeks
  Forced vital capacity (FVC), is the maximum amount of air that can be exhaled when blowing out as fast as possible. The pulmonary function test was evaluated with two different measurements, both at the beginning of the treatment (T0) and at the 8th week of the treatment (T1). The data obtained was determined as the primary outcome of the study, and the patients in both groups were administered by the research physiotherapist. For respiratory function tests were used a handheld type spirometer (SP10W, Contec). For the spirometric measurement, the patient was seated on the chair and a clip was placed on the patient nose to keep the nostril closed. Afterward, the device was placed in the patient's mouth, they were asked to take a deep breath and exhale into the device with maximum force. This process was repeated three times and the highest value among the measurements was recorded as respiratory function data.
FEV1 - Respiratory Functions | 8 Weeks
  Forced expiratory volume in 1 second (FEV1) is the volume of air exhaled in the first second during forced exhalation after maximum inspiration. The pulmonary function test was evaluated with two different measurements, both at the beginning of the treatment (T0) and at the 8th (T1) week of the treatment. The obtained data were determined as the primary outcome of the study and the patients in both groups were administered the same procedure by the researcher physiotherapist.
PEF - Respiratory Functions | 8 Weeks
  Peak expiratory flow (PEF), the maximal flow that can be exhaled when blowing out at a steady rate. The pulmonary function test was evaluated with two different measurements, both at the beginning of the treatment (T0) and at the 8th (T1) week of the treatment. The obtained data were determined as the primary outcome of the study and the patients in both groups were administered the same procedure by the researcher physiotherapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No